CLINICAL TRIAL: NCT05228704
Title: Study on the Influence of Forest Therapy on Healing Experience in Botanical Gardens.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Chung-Hua Hsu, Clinical Professor, Taipei City Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: TCHIRB-11002014
Record Dates: First submitted 2021-12-08; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Nature, Human
Keywords: Forest therapy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- activities in the Botanical Garden or Urban (Experimental): experiment group is activities in the Botanical Garden, and the control group is activities in urban
  Interventions: Behavioral: activities in the Botanical Garden or in urban
- Cross-over design (Other): The participants are randomized divided into in two groups following by the experiment which is designed by two consecutive times at one week intervals, and the experimental activities and the control activities are staggered.
  Interventions: Behavioral: activities in the Botanical Garden or in urban

INTERVENTIONS:
Behavioral: activities in the Botanical Garden or in urban — activities in the Taipei Botanical Garden or in Urban

SUMMARY:
The forest healing system is an important topic of alternative therapy in recent years. To study the influence of Forest therapy, the establishment of a pilot experimental model system in which both environmental factors and type of activity are necessary. Therefore, a system based on the Taipei Botanical Garden was introduced by this study.

DETAILED DESCRIPTION:
The forest healing system is an important topic of alternative therapy in recent years. Forest therapy began in 1989 when the psychology professor Kaplan put forward the "Attention Restoration Theory(ART)". Awareness has a positive benefit. To study the influence of Forest therapy, the establishment of a pilot experimental model system in which both environmental factors and type of activity are controlled can greatly reduce the errors caused by the site and the content of the activity. Therefore, a randomized controlled crossover experiment based on the Taipei Botanical Garden was introduced by this study.

ELIGIBILITY:
Inclusion Criteria:

* 20-35 years old youth (not limited to men and women)
* Those who have the ability and physical strength to walk for more than 120 minutes
* Subjects must voluntarily join the study

Exclusion Criteria:

* People who smoke or chew betel nuts
* People who have the habit of drinking (drinking more than five standard glasses in any situation)
* Drug addiction (including narcotic drugs and non-narcotics) habitual
* Those who have taken psychosomatic drugs in the past 30 days
* Participating in another clinical trial at the same time, or in the follow-up period of an interventional trial
* Those diagnosed with major injuries
* Women who are currently pregnant or breastfeeding
* Conditions where other subjects cannot cooperate (for example: unable to participate after random assignment, and not signing the subject's consent form)

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
questionnaire: BPOMS (1st) | baseline, pre-intervention(1st) → 2 hours intervention → immediately after the intervention(1st)
  Change from baseline Brief Profile of Mood States at first intervention
questionnaire: BPOMS (2nd) | pre-intervention(2nd) → 2 hours intervention → immediately after the intervention(2nd)
  Change from Brief Profile of Mood States at second intervention after 7-day-washout period & cross-over
questionnaire: BAI (1st) | baseline, pre-intervention(1st) → 2 hours intervention → immediately after the intervention(1st)
  Change from baseline The Beck Anxiety Inventory at first intervention
questionnaire: BAI (2nd) | pre-intervention(2nd) → 2 hours intervention → immediately after the intervention(2nd)
  Change from The Beck Anxiety Inventory at second intervention after 7-day-washout
questionnaire: BDI-II (1st) | baseline, pre-intervention(1st) → 2 hours intervention → immediately after the intervention(1st)
  Change from baseline The Beck Depression Inventory II at first intervention
questionnaire: BDI-II (2nd) | pre-intervention(2nd) → 2 hours intervention → immediately after the intervention(2nd)
  Change from The Beck Depression Inventory II at second intervention after 7-day-washout
questionnaire: BSRS-V (1st) | baseline, pre-intervention(1st) → 2 hours intervention → immediately after the intervention(1st)
  Change from baseline Brief Symptom Rating Scale V at first intervention
questionnaire: BSRS-V (2nd) | pre-intervention(2nd) → 2 hours intervention → immediately after the intervention(2nd)
  Change from Brief Symptom Rating Scale V at second intervention after 7-day-washout
physiological indicator: alpha-amylase activity in salivary (1st) | baseline, pre-intervention(1st) → 2 hours intervention → immediately after the intervention(1st)
  Change from baseline alpha-amylase activity in salivary by using commercial kits (Salimetrics®) at first intervention
physiological indicator: alpha-amylase activity in salivary (2nd) | pre-intervention(2nd) → 2 hours intervention → immediately after the intervention(2nd)
  Change from alpha-amylase activity in salivary by using commercial kits (Salimetrics®) at second intervention after 7-day-washout
physiological indicator: HRV (Heart Rate Variability) (1st) | baseline, pre-intervention(1st) → 2 hours intervention → immediately after the intervention(1st)
  Change from baseline HRV by using wrist monitors (ANSWatch®) to measure heart rate, heart rate variability (related to activities of the autonomic nervous system ANS), irregular heartbeats (IRRHB), and 5-minute continuous pulse wave at first intervention
physiological indicator: HRV (Heart Rate Variability) (2nd) | pre-intervention(2nd) → 2 hours intervention → immediately after the intervention(2nd)
  Change from HRV by using wrist monitors (ANSWatch®) to measure heart rate, heart rate variability (related to activities of the autonomic nervous system ANS), irregular heartbeats (IRRHB), and 5-minute continuous pulse wave at second intervention after 7-day-washout
physiological indicator: blood pressures (systolic and diastolic) (1st) | baseline, pre-intervention(1st) → 2 hours intervention → immediately after the intervention(1st)
  Change from baseline blood pressures by using wrist monitors (ANSWatch®) to measure blood pressures (systolic and diastolic) at first intervention
physiological indicator: blood pressures (systolic and diastolic) (2nd) | pre-intervention(2nd) → 2 hours intervention → immediately after the intervention(2nd)
  Change from blood pressures by using wrist monitors (ANSWatch®) to measure blood pressures (systolic and diastolic) at second intervention after 7-day-washout

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Hua Hsu, Study Director — Branch of Chinese Medicine, Taipei City Hospital
Locations (1):
- Taipei city hospital, Taipei, Taiwan